CLINICAL TRIAL: NCT05526521
Title: A Multi-center, Single-arm Study to Investigate the Pharmacokinetics and Safety of Dupilumab in Male and Female Participants ≥2 Years to <12 Years of Age With Uncontrolled Chronic Spontaneous Urticaria (CSU)
Brief Title: A Study to Investigate the Pharmacokinetics and Safety of Dupilumab in Participants ≥2 Years to <12 Years of Age With Uncontrolled Chronic Spontaneous Urticaria (CSU) (LIBERTY-CSU CUPIDKids)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKM16982; U1111-1266-5669 (Registry Identifier: ICTRP); 2022-000260-22 (EudraCT Number)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Administered subcutaneously (SC) every 4 weeks (Q4W) or every 2 weeks (Q2W) with or without an initial loading dose based on weight and age
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Injection solution Subcutaneous
  Other Names: Dupixent

SUMMARY:
This was a multicenter, single-arm, 24-week treatment, Phase 3 study. The purpose of this study was to investigate the PK and safety of dupilumab in children diagnosed with CSU who remain symptomatic despite the use of H1-antihistamine treatment. Study details included: Screening: 2 to 4 weeks; The treatment duration was 24 weeks; Follow-up period: 12 weeks; The study duration was 38 to 40 weeks (including screening and follow-up); The number of study visits was 6.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 2 years to <12 years of age, at the time of signing the informed consent.
* Participants who had history of a diagnosis of CSU prior to screening (Visit 1) or symptoms consistent with a diagnosis of CSU for at least 3 months in the Investigator's opinion.
* Participants with CSU (characterized by recurrent itchy wheals with or without angioedema for >6 weeks) who remain symptomatic at the time of screening despite regular H1-antihistamine treatment.
* Body weight within ≥5 kg to <60 kg.
* Participant/parent(s)/caregiver(s)/participant's legally authorized representative, as appropriate, willing and able to comply with study visits and related procedures.

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria apply:

* Underlying etiology for chronic urticarias other than CSU.
* Presence of skin morbidities other than CSU that may interfere with the assessment of the study outcomes.
* Participants with a diagnosis of chronic inducible cold urticaria.
* Participants with active AD.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study.
* Participants with active tuberculosis (TB) or non-tuberculous mycobacterial infection, or a history of incompletely treated.
* Diagnosed with, suspected of, or at high risk of endoparasitic infection.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the screening visit or during the screening period.
* Known or suspected immunodeficiency.
* Active malignancy or history of malignancy within 5 years before the baseline visit.
* History of systemic hypersensitivity or anaphylaxis to dupilumab including any excipient.
* Participation in prior dupilumab clinical study or have been treated with commercially available dupilumab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (9):
  - Pediatric Dermatology of Miami Site Number : 8400015, Coral Gables, Florida
  - Treasure Valley Medical Research Site Number : 8400019, Boise, Idaho
  - Washington University School of Medicine- Site Number : 8400004, St Louis, Missouri
  - Boston Childrens Health Physicians Site Number : 8400017, Hawthorne, New York
  - Columbia University Irving Medical Center Site Number : 8400003, New York, New York
  - Childrens Hospital Medical Center of Akron- Site Number : 8400020, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center - PIN- Site Number : 8400001, Cincinnati, Ohio
  - Vital Prospects Clinical Research Institute, P.C.- Site Number : 8400002, Tulsa, Oklahoma
  - Monroe Carell Jr. Childrens Hospital at Vanderbilt- Site Number : 8400005, Nashville, Tennessee
- Canada (4):
  - Investigational Site Number : 1240009, Calgary, Alberta
  - Investigational Site Number : 1240010, Edmonton, Alberta
  - Investigational Site Number : 1240007, Hamilton, Ontario
  - Investigational Site Number : 1240001, Montreal, Quebec
- Japan (2):
  - Investigational Site Number : 3920001, Yokohama, Kanagawa
  - Investigational Site Number : 3920002, Tsu, Mie-ken

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM16982 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25324&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 sites in Canada, Japan and the United States. A total of 23 participants were screened from 25-Aug-2022 to 02-May-2024 of which 8 were screen failures mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 15 participants were enrolled in the study to receive dupilumab at 1 of 4 dose regimens based on the body weight and age.
Groups:
- Dupilumab 200 mg Q4W: Participants received dupilumab 200 milligrams (mg) subcutaneous (SC) injection every 4 weeks (Q4W) with no loading dose in children aged >=2 years to <12 years with body weight >=5 kilograms (kg) and <15 kg from Day 1 up to 24 weeks.
- Dupilumab 300 mg Q4W: Participants received dupilumab 300 mg SC injection Q4W with no loading dose in children aged >=2 years to <6 years with body weight >=15 kg and <30 kg from Day 1 up to 24 weeks.
- Dupilumab 300 mg Q4W, 600 mg Loading Dose: Participants received dupilumab 300 mg SC injection Q4W with an initial 600 mg loading dose in children aged >=6 years to <12 years with body weight >=15 kg and <30 kg from Day 1 up to 24 weeks.
- Dupilumab 200 mg Q2W, 400 mg Loading Dose: Participants received dupilumab 200 mg SC injection every 2 weeks (Q2W) with an initial 400 mg loading dose in children aged >=2 years to <12 years with body weight >=30 kg and <60 kg from Day 1 up to 24 weeks.
Period: Overall Study
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Started | 1 | 4 | 2 | 8
Completed | 1 | 3 | 2 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who took at least 1 dose of the study intervention, regardless of the amount of intervention administered.
Groups:
- Dupilumab 200 mg Q4W: Participants received dupilumab 200 mg SC injection Q4W with no loading dose in children aged >=2 years to <12 years with body weight >=5 kg and <15 kg from Day 1 up to 24 weeks.
- Dupilumab 200 mg Q2W, 400 mg Loading Dose: Participants received dupilumab 200 mg SC injection Q2W with an initial 400 mg loading dose in children aged >=2 years to <12 years with body weight >=30 kg and <60 kg from Day 1 up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose | Total
Number analyzed (Participants) | 1 | 4 | 2 | 8 | 15
Age, Customized [Count of Participants; unit: Participants]
  >=2 to <6 years | 0 | 4 | 0 | 0 | 4
  >=6 to <12 years | 1 | 0 | 2 | 8 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 6 | 11
  Male | 0 | 2 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 0 | 4 | 1 | 4 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentration of Dupilumab at Weeks 12 and 24
Description: Blood samples were collected at specified timepoints to obtain dupilumab concentration.
Time Frame: Weeks 12 and 24
Population: The pharmacokinetic (PK) population included all enrolled and treated participants (safety population) with at least 1 post-baseline PK result. Only those participants with data collected at Weeks 12 or 24 are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 3 | 2 | 8
nanogram/milliliter
  Week 12: number analyzed (Participants) | 1 | 1 | 2 | 8
  Week 12 | 67700 | 105000 | 45800 (12400) | 91600 (23000)
  Week 24 | 116000 | 141000 (30100) | 51100 (20100) | 78500 (31600)

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of study intervention, whether or not considered related to study intervention. Serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From the first dose of study intervention (Day 1) up to end of follow-up, maximum up to 36 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 4 | 2 | 8
Participants
  TEAEs | 1 | 2 | 2 | 7
  TESAEs | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) to Dupilumab
Description: Blood samples were collected at specified timepoints and ADA samples were assayed using validated methods. Treatment-emergent ADA response was defined as a positive response in the ADA assay post first dose when baseline results were negative or missing. Number of participants with treatment-emergent ADA response is presented.
Time Frame: From the first dose of study intervention (Day 1) up to end of follow-up, maximum up to 36 weeks
Population: The ADA population included all enrolled participants treated with dupilumab with at least 1 post-baseline ADA result (positive, negative or inconclusive).
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 3 | 2 | 8
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (C-DLQI) in Participants Aged 4 Years to <12 Years at Week 24
Description: The C-DLQI assesses impact of skin disease on children's health-related quality of life (HRQoL) over the previous week, contains 10 questions related to symptoms feelings associated with disease, impact of disease on leisure, school or holidays, personal relationships, sleep, and side effects of treatment for the skin disease. All questions were scored on 4-point Likert scale:0 (not at all),1 (a little),2 (a lot),3 (very much). Total C-DLQI was calculated by summing the score of each question and ranged from 0 (no impact) to 30 (severe impact). Higher scores indicated poor HRQoL. Mean is presented. Baseline was defined as closest assessment to first study intervention administration on or prior to Day 1 but no later than Day 4.
Time Frame: Baseline (Day 1) and Week 24
Population: The intent-to-treat (ITT) population included all enrolled participants. Only those participants with data collected at Baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 1 | 2 | 7
score on a scale | -3.0 | -6.0 | -10.5 (3.5) | -7.3 (4.3)

5. Secondary Outcome: Change From Baseline in Infant's Dermatitis Quality of Life Index (IDQOL) in Participants Aged 2 Years to <4 Years at Week 24
Description: The IDQOL questionnaire is completed by child's caregiver/guardian with a recall period of 7 days;consists of 10 questions focusing on life quality index (LQI) scored on 4-point Likert scale. An additional question on dermatitis severity is scored on a 5-point Likert scale (0 [none] to 4 [extremely severe]); it is not considered for calculating total IDQOL. For LQI, score ranges are as follows: Questions 1, 5 to 10: 0 (none) to 3 (all the time/very much). Question 2: 0 (happy), 1 (slightly fretful), 2 (very fretful),3 (always crying). Question 3: 0 (0-15 minutes), 1 (15 minutes-1 hour), 2 (1-2 hours),3 (>2 hours).Question 4: 0 (<1 hour), 1 (1-2 hours), 2 (3-4 hours),3 (>=5 hours). IDQOL total score is the sum of the score of each question of LQI, ranges from 0 (no impact) to 30 (maximum impact). Higher scores indicated poor HRQoL. Mean is presented. Baseline was defined as closest assessment to first study intervention administration on or prior to Day 1 but no later than Day 4.
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT population included all enrolled participants. Only those participants with data collected at Baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 0 | 1 | 0 | 0
score on a scale |  | -3.0 |  |

6. Secondary Outcome: Change From Baseline in Modified Urticaria Activity Score Over 7 Days (mUAS7) at Week 24
Description: A modified version of the UAS (mUAS) was used for the smaller body surface area of child and adolescent participants. The mUAS was derived from the sum of daily hives severity score (HSS) (ranging from 0 to 3 [0 = absent; 1 = mild {1 to <10 wheals/24 hours}; 2 = moderate: {10 to 30 wheals/24 hours}; and 3 = intense: {>30 wheals/24 hours or large confluent areas of wheals}]) and daily itch severity score (ISS) (ranging from 0 = none to 3 = intense). Daily mUAS total scores range from 0 to 6 (0 to 3 for ISS and 0 to 3 for HSS). Daily mUAS scores were summed over 7-day period to create total score ranging from 0 (no urticaria) to 42 (severe urticaria). Completion of mUAS7 was done by the child or parent(s)/caregiver(s)/legal guardian(s) for participants aged >=4 years and by parent(s)/caregiver(s) for participants aged <4 years. Mean is presented. Baseline was defined as sum of the 7 daily measurements obtained within the 7 days prior to first study intervention administration.
Time Frame: Baseline (Day -7 to Day 1) and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 2 | 2 | 5
score on a scale | -8.0 | -21.4 (1.9) | -2.8 (1.8) | -7.8 (6.6)

7. Secondary Outcome: Change From Baseline in Itch Severity Score Over 7 Days (ISS7) at Week 24
Description: The ISS represents severity of itch on a scale ranging from 0 (none) to 3 (intense). The ISS7 score was the sum of daily ISS scores recorded by a participant at the same time each day over 7 days with an overall scale of 0 (no impact) to 21 (severe impact). Higher scores indicated greater intensity of itch. Mean is presented. Baseline was defined as sum of the 7 daily measurements obtained within the 7 days prior to first study intervention administration.
Time Frame: Baseline (Day -7 to Day 1) and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 2 | 2 | 5
score on a scale | -5.0 | -9.6 (3.7) | -1.6 (0.6) | -3.4 (3.2)

8. Secondary Outcome: Change From Baseline in Hive Severity Score Over 7 Days (HSS7) at Week 24
Description: The HSS7 score is the sum of daily HSS ranging from ranging from 0 to 3 (0 = absent; 1 = mild [1 to <10 wheals/24 hours]; 2 = moderate [10 to 30 wheals/24 hours]; and 3 = intense: [>30 wheals/24 hours or large confluent areas of wheals]) recorded by a participant at the same time of each day over 7 days with an overall scale of 0 (no hives) to 21 (severe hives). Higher scores indicate greater intensity of hives. Mean is presented. Baseline was defined as sum of the 7 daily measurements obtained within the 7 days prior to first study intervention administration.
Time Frame: Baseline (Day -7 to Day 1) and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
Number analyzed (Participants) | 1 | 2 | 2 | 5
score on a scale | -3.0 | -11.8 (1.8) | -1.2 (1.2) | -4.4 (3.6)

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention (Day 1) up to end of follow-up, maximum up to 36 weeks
Description: Analysis was performed on the safety population.
Arm/Group | Dupilumab 200 mg Q4W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q4W, 600 mg Loading Dose | Dupilumab 200 mg Q2W, 400 mg Loading Dose
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 1/1 | 2/4 | 2/2 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab 200 mg Q4W (N=1) | Dupilumab 300 mg Q4W (N=4) | Dupilumab 300 mg Q4W, 600 mg Loading Dose (N=2) | Dupilumab 200 mg Q2W, 400 mg Loading Dose (N=8)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral Rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Internal Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling Face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT05526521/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT05526521/SAP_001.pdf